CLINICAL TRIAL: NCT06254248
Title: Safety of Atezolizumab-Bevacizumab in Liver Transplanted Patients With Advanced Hepatocellular Carcinoma
Acronym: IMMUNO-TH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230899
Record Dates: First submitted 2024-01-12; First posted 2024-02-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplant; Hepatocellular Carcinoma Recurrent; Systemic Treatment
Keywords: HCC; systemic therapy; graft rejection; immunotherapy; Atezolizumab-Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezo-Beva combination (Experimental): first-line Atezo-Beva combination in LT patients with advanced HCC in association with a standardized immunosuppressive treatment to prevent the risk of acute cellular rejection
  Interventions: Drug: Systemic therapy

INTERVENTIONS:
Drug: Systemic therapy — Atezolizumab-Bevacizumab every 3 weeks until progression or side effects in combination with Standardized immunosuppressive treatment:
  Tacrolimus (objective 5-7 ng/ml) Mycophenolate Mofetil 1000 mg per day Corticosteroids at least 5 mg per day Everolimus will be continued if already started before the inclusion (objective 5-7 ng/ml). If everolimus has not been started prior to inclusion, do not start it, but adopt the following protocol: corticoids + Tacrolimus + Cellcept.

SUMMARY:
The prognosis of liver transplanted (LT) patients with recurrence of hepatocellular carcinoma (HCC), especially those with progression after locoregional treatment or advanced HCC, remains poor. Current treatment modalities involve tyrosine kinase inhibitors (TKIs) characterized by a low response rate and often poor tolerability. Encouraging findings from the Imbrave 150 study, demonstrating increased survival rates coupled with favorable treatment tolerance, prompt the investigators to consider the potential of offering the combination of treatment with Atezolizumab-Bevacizumab (Atezo-Beva) to patients with LT. No data regarding the safety and efficacy of this new combination are available for patients with LT as they were not included in Imbrave 150. Immunosuppression after LT is low when compared to essentially all other organ recipients, liver recipients are considered with lower immunological risk. However, the use of ICIs has been associated with a risk of hepatic rejection in LT patients. In this study, in order to prevent acute cellular rejection (ACR) occurrence, we propose to adopt a standardized immunosuppressive regimen closed to the one used immediately after LT but with lower therapeutic goals for tacrolimus and everolimus to allow immunotherapy treatment to be effective. The better tolerance of liver grafts will probably lead to less risk of rejection with Atezo-Beva than in other organ transplants.

DETAILED DESCRIPTION:
Open-label multicentric single-arm two-stage phase 2 trial. Population: Adult LT patients with advanced HCC recurrence with indication to systemic treatment Primary objective: To study the safety (ACR on histology) at 6 months of the first-line Atezo-Beva combination in LT patients with recurrent HCC in association with a standardized immunosuppressive treatment to prevent the risk of liver graft rejection.

Primary endpoint: Rate of Acute cellular rejection (ACR) (defined by a Histological Banff score ≥ 5) at 6 months (confirmed by an external expert center).

Secondary objective:

To study the safety (ACR on histology) at 24 months and at the end of Atezo-Beva treatment in LT patients with recurrent HCC in association with a standardized immunosuppressive treatment to prevent the risk of liver graft rejection.

* To assess the efficacy and tolerance of first-line Atezo-Beva combination in LT patients with advanced HCC in association with a standardized immunosuppressive treatment to prevent the risk of ACR based on:
* the Progression Free Survival (PFS)
* the Overall survival (OS)
* the objective response rate (ORR) (complete and partial response)
* the duration of response
* the quality of life of the patients under Atezo-Beva treatment
* To compare the efficacy (OS and PFS) of LT patients treated by Atezo- Beva treatment to an historical retrospective cohort of LT patients already available treated by TKI as first line (external arm comparison)
* To assess the adverse events related to Atezo-Beva treatment in LT patients with recurrent advanced HCC.
* To assess the evolution of the level of donor specific antibodies (DSA) during Atezo-Beva treatment and its association with ACR, PFS and OS.

Translational research/ancillary studies:

* To assess the association before the first injection between the risk of ACR, PFS, OS and side effects and
* the "Immunome" imaging on tumor sample and non-tumoral liver sample to quantify and regionalize immune populations on pathology (Multispectral Imaging, Mantra)
* the Leukocyte DNA analysis to identify constitutional genetic variants
* To assess the association before the first injection or just before the second injection and at 3 months between the risk of ACR, PFS, OS and side effects and
* the "immunomonitoring" on blood sample (frequency and/or the phenotype of circulating immune cells)
* the presence of tumors cells (liquid biopsies)
* the presence of circulating tumor DNA and the type of mutations
* the presence of circulating proteins
* the profile of circulating exosomes

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 and under 90 years old:
* who underwent LT more than 6 months ago (to prevent the higher risk of ACR which exists within the first months after LT and to deal with populations with a lowered immunosuppressive regimen long after LT)
* with HCC recurrence diagnosis according to the EASL diagnostic criteria (33)
* with advanced HCC not accessible to surgery and locoregional treatment
* with at least one measurable untreated lesion
* With a proposal for Atezo-Beva in first line treatment made in a multidisciplinary meeting
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment, unless otherwise specified:

  * ANC ≥ 1.5 x 109/L (1500/µL) without granulocyte colony-stimulating factor support
  * Lymphocyte count ≥ 0.5 x 109/L (500/µL)
  * Platelet count ≥ 75 x 109/L (75,000/µL) without transfusion
  * Hemoglobin ≥ 90 g/L (9 g/dL). Patients may be transfused to meet this criterion.
  * AST, ALT ≤ 5 x upper limit of normal (ULN)
  * Serum bilirubin ≤ 3x ULN
  * creatinine clearance≥40 mL/min (calculated using the Cockcroft-Gault formula)
  * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 2x ULN
  * Urine dipstick for proteinuria < 2+ (within 7 days prior to initiation of study treatment). Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1 g of protein in 24 hours
* ECOG Performance Status of 0 or 1
* For women of childbearing potential and men: agreement to remain abstinent or use effective contraception during treatment and at least :

  * 5 months after the end of the treatment with atezolizumab,
  * 6 months after the end of the treatment with bevacizumab
* Child-Pugh class A

Exclusion Criteria:

* History of ACR within 3 months before starting Atezo-Beva treatment
* Banff score for ACR ≥ 3 on liver biopsy performed before the initiation of the treatment
* Pregnant or breastfeeding woman
* Patient not affiliated to a beneficiary or entitled social security scheme or to the PUMA
* Patient not having signed consent
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT-scan
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) ≥ 160 mmHg and/or diastolic blood pressure > 100 mmHg), based on an average of ≥ 3 BP readings on ≥ 2 sessions Anti-hypertensive therapy to achieve these parameters is allowable.
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses
* Hypersensitivity to the active substance or to any of the excipients of the SmPC of bevacizumab and the SmPC of atezolizumab
* Hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies
* Prior arterial thromboembolic reactions including cerebrovascular accidents, transient ischaemic attacks and myocardial infarctions;
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* In case of proteinuria > 1g in 24 hours
* History of leptomeningeal disease
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Acute cellular rejection (ACR) (defined by a Histological Banff score ≥ 5) at 6 months (confirmed by an external expert center) | 6 months
  To study the safety (ACR on histology) at 6 months of the first-line Atezo-Beva combination in LT patients with recurrent HCC in association with a standardized immunosuppressive treatment to prevent the risk of liver graft rejection

SECONDARY OUTCOMES:
Rate of Acute Cellular Rejection (ACR) at 24 months | 24 months
  Rate of ACR (defined by a Histological Banff score ≥ 5) at 24 months (confirmed by a second external expert center.
Rate of Acute Cellular Rejection (ACR) at the end of Atezo-Beva treatment | at the end of treatment
  Rate of ACR (defined by a Histological Banff score ≥ 5) at 24 months and at the end of Atezo-Beva treatment (confirmed by a second external expert center.
Progression Free Survival (PFS) | between the inclusion and 24 months after the last inclusion
  The Progression Free Survival (PFS) is defined as the time from inclusion to disease progression according to RECIST 1.1 on imaging (CT-scan) performed every 3 months or death from any cause, whichever occurred first.
Overall survival (OS) | between the inclusion and 24 months after the last inclusion
  The Overall survival (OS) defined by the time from inclusion to death from any cause
Objective Response Rate (ORR) | 12 months
  The Objective Response Rate (ORR) at 12 months is defined as the percentage of patients with a confirmed complete or partial response according to RECIST 1.1 criteria on imaging (CT-scan) performed every 3 months.
Duration of response | between the inclusion and 24 months after the last inclusion
  The Duration of response is defined by the time from first documentation of complete or partial response to disease progression or death according to RECIST 1.1 criteria on imaging (CT-scan) performed every 3 months.
Time to deterioration of quality of life | between the inclusion and 24 months after the last inclusion
  The time to deterioration of quality of life is defined as the time from inclusion to the first deterioration of quality of life as reported by the patient, with deterioration defined as a decrease from baseline of 10 points or more on the EORTC QLQ-C30 maintained for two consecutive assessments or a decrease of 10 points or more in one assessment followed by death from any cause within 3 weeks. Each quality of life evaluation will be reported by the patient using EORTC QLQ-C30 score fill formed every 6 months until 24 months after the initiation of the treatment.
Type, frequency and severity of adverse events and serious adverse events | between the inclusion, at the end of Atezo-Bev treatment and up to 24 months
  They will be assessed on the basis of the nature, frequency and severity of adverse events according to NCI Common Terminology Criteria for Adverse Events, version 4.0. The management of side effects usually observed under immunotherapy will be managed according to the American Society of Clinical Oncology Clinical Practice Guidelines
Donor Specific Antibodies (DSA) median | baseline and at Day 21, 3 Months 6 Months , 12 Months , 18 Months , 24 Months
  DSA will be assessed and correlation to ACR, the PFS and OS will be evaluated

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Hôpital Beaujon, Clichy
  - Hôpital Henri-Mondor, Créteil
  - Hôpital Claude Huriez - CHU de Lille, Lille
  - Lyon - Hôpital Croix Rousse, Lyon
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - Hôpital de Hautepierre - Strasbourg, Strasbourg
  - CHU Tours - Hôpital Trousseau, Tours
  - Hôpital Paul Brousse, Villejuif